CLINICAL TRIAL: NCT06632535
Title: Group Medical Visits and Chiropractic Care for Older Adults With Chronic Spine Pain
Acronym: GOLDEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter M. Wayne, Ph.D., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002528
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: chiropractic; group medical visit; shared medical visit; older adults; spine pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined chiropractic care and group medical visits (Experimental): Participants will attend 8 weekly chiropractic visits (40-minutes for initial visit, 20-minutes for remaining 7). Participants will simultaneously enroll in 8 weekly 90-minute virtual group medical visits.
  Interventions: Other: Chiropractic care; Other: Group medical visits

INTERVENTIONS:
Other: Chiropractic care — Chiropractic treatment will involve a personalized treatment plan within the context of a general care protocol administered by a chiropractor at the Osher Clinical Center for Integrative Health. The treatment plan will be customized to the patient's clinical needs following the current evidence and clinical practice guidelines.
Other: Group medical visits — Participants will simultaneously enroll in virtual group medical visits with group discussion, practice based learning, and curricular themes pertaining to chronic pain management, healthy aging, and pillars of lifestyle medicine.

SUMMARY:
Chronic spine pain is one of the most common and conditions in adults over the age of 65. Treatments for pain that are non-pharmacologic (do not use over-the-counter or prescription drugs) are recognized as some of the most important to study. Chiropractic care has shown to be effective at reducing chronic pain, and growing research supports the use of group visit programs for the management of chronic pain. There is reason to believe that combining the two could enhance the benefit previously demonstrated by these treatments individually. There are no studies that have examined the combined delivery of chiropractic care and group visit programs for adults over the age of 65. The investigators plan assess the feasibility of treating adults over the age of 65 with chronic spine pain with chiropractic care and a group visit program. A battery of biopsychosocial outcomes will be collected to inform a more definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years of age
* Chronic neck, thoracic, and/or low back pain at least 5 days a week for at least 3 consecutive months
* Neck, thoracic, and/or low back pain averaged over past week of 3 or more on numerical rating scale ranging from 0 to 10, with 10 described as 'worst pain imaginable'
* Oswestry Disability Index score of 10% or greater
* Access to and ability to use a smartphone, tablet, or computer and broadband internet
* Access to reliable mode of transportation for study visits and chiropractic treatments
* Agreeable to participate in all study procedures
* Fluent in English

Exclusion Criteria:

* Currently, or having received chiropractic care in past 12 months (for any spine pain condition)
* Any disability precluding safe exercise practice
* Any prior spinal surgery within previous year
* Persons currently involved in a disability/accident claim
* Currently living in a nursing home and/or enrolled in hospice
* Need for additional diagnostic imaging at the eligibility exam
* Signs/symptoms of major systemic illness that may impair the participant's ability to effectively attend intervention sessions, or present risk factors to the care protocol: Participants with signs or symptoms suggesting the need for evaluation and/or management by other providers (e.g., Parkinson's disease, cancer, psychosis, substance use addiction)
* Non-neuromusculoskeletal source: Participants with neck or back pain suspected or confirmed non-neuromusculoskeletal source (e.g., vasculitis, referred pain of cardiopulmonary origin, neoplasm, or infection)
* Inflammatory arthritis: Participants suspected or confirmed diagnosis of rheumatoid arthritis, ankylosing spondylitis or other systemic inflammatory arthritis condition
* Health conditions influencing compliance: Participants with health conditions that lead to difficulty complying with study protocol, such as renal dialysis, untreated psychiatric symptoms, or cognitive impairment
* Vascular risk: Participants at increased risk for adverse cerebrovascular events are ineligible. Examples include a history of stroke, carotid artery dissection, or vertebral artery dissection, and those scheduled for endarterectomy procedures due to arterial stenosis. The presence of carotid artery bruit is exclusionary due to a presumed increased vascular risk and the likely need for referral and diagnostic testing
* Neurological disorder: Participants exhibiting a clinical picture of serious or potentially serious neurological disorders are ineligible. Examples include:

  * Progressive neurologic deficit evidenced by signs/symptoms such as paralysis, progressive muscle weakness, poor coordination, loss of sensation, and loss of bladder or bowel function
  * Suspected or confirmed myelopathy or radiculopathy
  * Space occupying lesions, within or adjacent to the spinal canal, including tumors (benign or malignant)
  * Neurological deficit (loss of sensation, motor strength, and/or deep tendon reflexes) present for less than 12 months

    * Note: The presence of a cervical disc herniation/protrusion is not exclusionary without signs of neurological deficit.
    * Note: Stable neurological deficit (present for more than 12 months without change) is not exclusionary
* Pathological hypermobility: Participants with suspected or confirmed diagnosis of a disorder known to cause spinal joint hypermobility including congenital conditions (Marfan Syndrome, Ehlers-Danlos Syndrome, and Osteogenesis imperfecta) and degenerative or traumatic instability are ineligible. Potential participants will be screened using Beighton criteria, health history, and (when available) diagnostic imaging review.
* Contraindication: Participants with confirmed or suspected contraindication to care not otherwise described (e.g., cervical fracture) are ineligible. This criterion does not include factors representing relative contraindications to specific procedures such as the presence of osteoporosis, for which chiropractic care can be safely adapted.
* Recent interventional pain management: defined as procedures such as corticosteroid injection, trigger point injection, and radiofrequency ablation to the cervical or lumbar region within the past 4 weeks and/or scheduled for interventional pain management procedures within the study timeframe.
* Hearing or visual impairment affecting participation in a virtual program

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Prior to intervention initiation
  Recruitment will be evaluated by tracking the recruitment source of participants, the number of participants enrolled per week overall, the reasons that screened individuals were not eligible, and the number of individuals deciding not to be screened, or if screened, why they are not interested in enrolling. Recruitment is estimated to be 10 total participants.
Retention | Monitored weekly throughout 8-week intervention period
  Retention will be quantified by the proportion of participants who complete all outcome assessments at the end of the intervention period. We will consider future testing of our interventions if the expected proportion of participants to have completed primary outcome assessments is least 70%.
Adherence | Monitored weekly throughout 8-week intervention period
  Adherence will be calculated as the proportion of participants who attend at least 6 of the 8 chiropractic care visits and 6 of the 8 of virtual group visits. We will consider future testing of our interventions if the expected proportion of participants judged to be adherent to the intervention is at least 70%.
Satisfaction with interventions | Measured at 8-week study visit
  Satisfaction will be calculated as the proportion of participants who report satisfaction with the program. We will consider future testing of our interventions if the expected proportion of participants who report satisfaction is at least 70%.

SECONDARY OUTCOMES:
Pain intensity | Measured at baseline and 8-week study visit
  Pain intensity will be measured using a 11-point numerical rating scale (NRS) with 0 indicating "no pain at all" and 10 indicating "worst pain imaginable".
Oswestry Disability Index | Measured at baseline and 8-week study visit
  Pain-related disability will be measured using the Oswestry Disability Index (ODI). These 10-item questionnaires determine how participants see their pain affecting their daily activities. The maximum score is 100%. Scores of <8% indicate no disability; 10% to 28% indicate mild disability, 30% to 48% moderate disability, and 50% to 68% severe disability. Scores >70% indicate a complete perceived disability.
PROMIS-29 | Measured at baseline and 8-week study visit
  PROMIS 29 is a system of validated, highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. In addition to pain intensity and pain interference, this set of measures includes physical function, fatigue, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.Raw scores are extracted and converted to T-scores on all subscales. Items are scored from 1 to 5, with a higher score indicating a higher degree of the construct being measured. The T-score metric used for data analysis uses a mean of 50 and a standard deviation of 10 in the U.S. population.
Self-efficacy | Measured at baseline and 8-week study visit
  Self-efficacy will be measured using the General Self-Efficacy Scale (GSES). The GSES measures a participant's confidence in their ability to respond to environmental demands and challenges. The scale consists of 10 items with a 4-point Likert response scale ranging from 1 ("not at all true") to 4 ("exactly true"). Higher summed scores indicate greater self-efficacy to complete tasks.
Locus of control | Measured at baseline and 8-week study visit
  Locus of control will be measured using the Internal-External Locus of Control short Scale-4 (IE-4). The IE-4 measures two dimensions of the locus of control (internal and external) with two items each. Each statement consists of a 5-point Likert scale with responses ranging from 1 ("doesn't apply at all") to 5 ("applies completely"). Higher scores in the first two items indicate an internal locus of control, while higher scores in the second two items indicate an external locus of control.
Pain catastrophizing | Measured at baseline and 8-week study visit
  Pain Catastrophizing Scale used to assess catastrophic thinking associated with pain. This instrument consists of 13 items that measure rumination, magnification, and helplessness related to pain and has adequate to excellent internal consistency, with higher scores representing more of the item tested.
Fear of Movement | Measured at baseline and 8-week study visit
  Fear of Movement will be measured using the Tampa Scale for Kinesiophobia. This instrument consists of 17 items that measure pain-related fear and has been validated in chronic low back pain and fibromyalgia patients. Higher scores represent more fear of movement.
Social Support | Measured at baseline and 8-week study visit
  Social Support will be measured with the Multidimensional Scale of Perceived Social Support (MSPSS) which measures an individual's perception of support from family, friends, and a significant other. It consists of 12 items with lower scores indicating low perceived support, and higher scores indicating higher perceived support.
Short Physical Performance Battery (SPPB) | Measured at baseline and 8-week study visit
  The SPPB measures lower extremity physical performance status including balance, gait speed, and chair stands and has been linked to mortality and disability. Gait speed, contained in the SPPB, will be assessed using the ZenoTM Walkway, developed by ProtoKinetics (https://www.protokinetics.com). The portable 2' X 20' gait walkway and associated hardware system can be easily assembled for use in a clinical setting (e.g., hallway), and comes with laptop computer with sophisticated, but user-friendly software (PKMAS). Gait data is collected by simply having the patient walk across an electronic gait mat. A series of gait parameters automatically calculated by ZENOTM will be captured including walking speed and stride time variability.
Qualitative interviews | Measured at baseline and 8-week study visit
  Qualitative interviews will be employed to further probe participants' perceptions of the combined interventions focusing on a) understanding facilitators and barriers to participation, and b) patient-centered experiences that might inform outcome measures to use in a future trial.

CONTACTS AND LOCATIONS:
Locations (1):
- MassGeneralBrigham, Boston, Massachusetts, United States